CLINICAL TRIAL: NCT02686840
Title: Sublingual Versus Vaginal Misoprostol In Medical Treatment of First Trimestric Missed Miscarriage: A Randomized Controlled Trial.
Brief Title: Sublingual Versus Vaginal Misoprostol In Medical Treatment of First Trimestric Missed Miscarriage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Abdel Shafy El Shahawy, Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASUMH
Record Dates: First submitted 2016-01-27; First posted 2016-02-22 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Missed Abortion
MeSH Terms: conditions — Abortion, Missed

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sublingual misoprostol (Experimental): Group A (100 patients): will be treated with sublingual misoprostol
  Interventions: Drug: sublingual misoprostol
- vaginal misoprostol (Active Comparator): Group B (100 patients): will be treated with vaginal misoprostol
  Interventions: Drug: vaginal misoprostol

INTERVENTIONS:
Drug: sublingual misoprostol — All patients will receive three doses of sublingual misoprostol every four hours The first dose of misoprostol 800 mcg will be administrated at the hospital. Then the patient will be observed for 1 hour for any immediate adverse reaction Clear instructions about the method and timing of second dose will be given upon sending home.
  * Two doses of misoprostol 800 mcg each (four tablets of 200 mcg per dose).
  * Paracetamol, eight hourly, will be provided as analgesic or antipyretic.
  * A specimen bottle to collect the POC if passed out.
  * Two pairs of disposable gloves.
  * Pre-filled histopathological examination form to be sent to the laboratory together with the products of conception
  Other Names: Misotac
  Arms: sublingual misoprostol
Drug: vaginal misoprostol — All patients will receive three doses of vaginal misoprostol every four hours The first dose of misoprostol 800 mcg will be administrated at the hospital. Then the patient will be observed for 1 hour for any immediate adverse reaction Clear instructions about the method and timing of second dose will be given upon sending home.
  Paracetamol, eight hourly, will be provided as analgesic or antipyretic
  Other Names: Misotac
  Arms: vaginal misoprostol

SUMMARY:
The aim of this work is to compare the effectiveness of vaginal versus sub-lingual misoprostol for medical treatment of first trimester missed miscarriage.

DETAILED DESCRIPTION:
In women with first trimetric-missed miscarriage, sublingual misoprostol may be as vaginal misoprostol in achievement of successful miscarriage so our aim was to compare the effectiveness of vaginal versus sub-lingual misoprostol for medical treatment of first trimester missed miscarriage.

ELIGIBILITY:
Inclusion Criteria:

* All women above 18 years of age
* Less than 12 weeks of gestation.
* Pregnancy is confirmed by pregnancy test or ultrasound scan.
* missed abortion
* Normal general and gynecological examination.
* The size of the uterus on pelvic examination was compatible with the estimated duration of pregnancy

Exclusion Criteria:

* Hemodynamically unstable.
* Suspected sepsis with temperature 38 °C.
* Concurrent medical illness e.g. hematological, cardiovascular, thromboembolism, respiratory illnesses, recent liver disease or pruritus of pregnancy.
* Presence of intrauterine contraceptive device (IUCD).
* Suspect or proven ectopic pregnancy.
* Failed medical or surgical evacuation before presentation.
* Known allergy to misoprostol.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Completeness of abortion: expulsion of Products of conception (POC)x by visual inspection | 7 days

SECONDARY OUTCOMES:
Successful medical abortion: cervical os is closed with endometrial thickness of less than 15 mm | 7 days
Failure: endometrial thickness of more than 15 mm on day seven (from third dose of misoprostol) or developing of complications before day seven needing early surgical evacuation. | 7 days
Bleeding pattern following treatment | 7 days
  This will be assessed by hemoglobin(g/dl) and haematocrit level after the treatment , if the patients required blood transfusion and number of units transfused and number of days of bleeding
Pain resulting from the procedure | 7 days
  this will be assessed by the doses of paracetamol given in mg
Additional uterotonic used | 7 days
  additional misoprostol doses in mcg

CONTACTS AND LOCATIONS:
Overall Officials: Hassan A Bayoumy, MD, Study Chair — Ain Shams University
Locations (1):
- Ain shams university maternity hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Abdelshafy A, Awwad H, Abo-Gamra A, Alanwar A, Elkotb AM, Shahin M, Abd El-Razek M, Abbas AM. Sublingual vs vaginal misoprostol for completion of first trimester missed abortion: a randomised controlled trial. Eur J Contracept Reprod Health Care. 2019 Apr;24(2):134-139. doi: 10.1080/13625187.2019.1569224. Epub 2019 Feb 12. PMID 30747547